CLINICAL TRIAL: NCT04772690
Title: Feasibility Study Exploring a Resource-orientered, Coordinated Rehabilitation and Palliative Care Intervention Among People With Advanced Cancer.
Brief Title: Balance, Activity and Quality of Life
Acronym: BAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REHPA
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAL (Experimental): A resource-orientered, individual and group-based intervention addressing balance in everyday life, activities and QoL among people with chronic or advanced cancer.
  Interventions: Other: A resource-oriented intervention

INTERVENTIONS:
Other: A resource-oriented intervention — The intervention is delivered by an interdisciplinary team of occupational therapist, physiotherapist, nurse, psychologist, physician and social worker. It consists of a five-day residential stay at REHPA and a two-day follow-up stay after seven weeks at home. The residential stays include both workshops and engagement in physical and creative activities.

SUMMARY:
Background: Advanced cancer may cause functional limitations, subsequently leading to decreased ability to perform and engage in everyday activities, such as self-care, household, leisure and civic life. In addition, people with advanced cancer need alleviation from the pain and sorrow following limited life expectancy wherefore they prefer to focus on everyday life function and activities, lightness and enjoyment. The overall aim of the Balance, Activity and quality of Life (BAL) project is to develop, test and evaluate effectiveness and process of a resource-oriented intervention which coordinates rehabilitation and palliative care to enhance quality of life (QoL), balance and enjoyment in everyday activities and functioning. The development of the intervention is guided by the British Medical Research Council's guidance (MRC).

The present study consists of a resource-oriented intervention, which will be feasibility tested in the research clinic of REHPA, the Danish Knowledge Centre for Rehabilitation and Palliative Care. The study will inform the development of a resource-oriented program for people with advanced cancer.

Material and Methods: A feasibility study designed as a one-armed, pre-post study with follow-up after five days and again after 6 and 12 weeks. The study will recruit 20-25 home-living adults (⩾18 years) with chronic or advanced cancer reporting needs in everyday life.

Outcomes are quality of life, physical function and fatigue assessed using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 (EORTC QLQ C-30). Furthermore, balance in everyday activities will be assessed using the Occupational Balance Questionnaire 11 (OBQ-11).

Besides outcomes, process data will also be collected regarding: 1) fidelity, 2) adherence, 3) dose and 4) reach and mechanisms of impact with attention to participant's experiences of and interactions with the intervention. These data will be collected using registration forms, questionnaires, participant-observations and focus-group interviews.

ELIGIBILITY:
Inclusion Criteria:

* Home-living adults
* Diagnosed with chronic or advanced cancer
* Report a need of support in everyday life and to better balance everyday life with necessary and meaningful activities
* Motivated and able to participate in the intervention
* Know sufficient Danish to complete questionnaires and participate in interviews

Exclusion Criteria:

* Dependent in basic activities of daily living (personal care, dressing and eating)
* Not able to complete questionnaires and participate in interviews
* Severe cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Change in global health status/ quality of life using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 | 6 week
  Scores between 0-100, with higher scores indicating better outcome

SECONDARY OUTCOMES:
Change in global health status/ quality of life using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 | 5 day
  Scores between 0-100, with higher scores indicating better outcome
Change in balance in everyday life using the Occupational Balance Questionnaire 11 | 5 day
  Scores between 11-44, with higher scores indicating better outcome
Change in physical function using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 | 5 day
  Scores between 0-100, with higher scores indicating better outcome
Change in fatigue using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 | 5 day
  Scores between 0-100, with higher scores indicating worse outcome
Change in balance in everyday life using the Occupational Balance Questionnaire 11 | 6 week
  Scores between 11-44, with higher scores indicating better outcome
Change in physical function using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 | 6 week
  Scores between 0-100, with higher scores indicating better outcome
Change in fatigue using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 | 6 week
  Scores between 0-100, with higher scores indicating worse outcome
Change in global health status/ quality of life using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 | 12 week
  Scores between 0-100, with higher scores indicating better outcome
Change in balance in everyday life using the Occupational Balance Questionnaire 11 | 12 week
  Scores between 11-44, with higher scores indicating better outcome
Change in physical function using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 | 12 week
  Scores between 0-100, with higher scores indicating better outcome
Change in fatigue using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 | 12 week
  Scores between 0-100, with higher scores indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sampedro Pilegaard, PhD, Principal Investigator — REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care; Karen la Cour, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- REHPA, the Danish Knowledge Centre for Rehabilitation and Palliative Care, Odense University Hospital, Nyborg, Denmark

REFERENCES:
- [Derived] Brunsgaard Laursen M, Sampedro Pilegaard M, la Cour K. Promising results of a resource- and activity-oriented intervention integrating rehabilitation into palliative care in people with advanced cancer: A feasibility study testing outcome measures. Palliat Support Care. 2025 Feb 7;23:e55. doi: 10.1017/S1478951524001652. PMID 39917823
- [Derived] Pilegaard MS, Timm H, Birkemose HK, Dupont SB, Joergensen DS, la Cour K. A resource-oriented intervention addressing balance in everyday activities and quality of life in people with advanced cancer: protocol for a feasibility study. Pilot Feasibility Stud. 2022 Apr 20;8(1):86. doi: 10.1186/s40814-022-01038-8. PMID 35443699